CLINICAL TRIAL: NCT03049670
Title: The Use of Klorsept Solution for Debriding Infected Wounds: is it Effective and Safe? Prospective Observational Study
Acronym: Klorsept
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Yaron Har-Shai, Clinical Professor of Plastic Surgery. Director, The Unit of Plastic Surgery, Carmel Medical Center
Other Study IDs: Any unique identifier assigned
Record Dates: First submitted 2017-01-15; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Non-healing Wound; Infected Wound
Keywords: Safety Issue
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- latent available chlorine (LAC): applying LAC on infected wounds
  Interventions: Device: latent available chlorine (LAC)

INTERVENTIONS:
Device: latent available chlorine (LAC) — local application on the necrotic infected tissue
  Other Names: K-sept

SUMMARY:
Klorsept is a debridement solution of necrotic infected tissue promoting wound healing. The aim of this study is to elaborate the effectiveness and safety of this solution.

DETAILED DESCRIPTION:
Klorsept is a debridement solution of necrotic infected tissue promoting wound healing. The aim of this study is to elaborate the effectiveness and safety of this solution.

This study will include 50 patients suffering from necrotic and infected wounds. Several parameters will be evaluated in order to provide the effectiveness and safety of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with infected wounds who can sign an informed consent

Exclusion Criteria:

* patient that can not sign an informed consent
* pregnant woman
* age less than 18 years
* Allergy to chlorine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females above the age of 18
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
antiseptic properties | 1 year
  General outcome: Pain will be assessed by the VAS scale. Score above 3 will be considered an abnormal value. Fever ( in C0) above 37.5 an abnormal value. Pulse rate elevated from the baseline patient by 15% will be an abnormal value. Systolic Blood pressure elevated from the baseline of the patient by 15% will be an abnormal value. Number of breathing which will be elevated from the baseline of the patient by 15% will be an abnormal value. Saturation which will be reduced by 5% from the baseline will be an abnormal value.
  Local Outcome: redness/ edema /odor/discharge will be evaluated by a score from 0 to 3 (0- no redness/edema/odor/discharge ; 3- severe redness /edema/odor/discharge). Skin eruption will be evaluated as no/yes.
  The results will be aggregated to arrive at one reported value (e.g., Number of Participants with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment)

SECONDARY OUTCOMES:
laboratory tests | 1 year
  laboratory tests: Glucose: values that are above 100 mg/dl (not with diabetic patients) Albumin: values that are less than 3.5 g/dl Creatinine: values that are above 1.17 mg% Urea: values that are above 43 mg% Sodium: values that are under 135 mEq/l or above 145 mEq/l Potassium: values that are under 3.5 mEq/l or above 5.1 mEq/l White blood count: values that are above 10.80 k/ul C- reactive protein: values that are above 0.5 mg/dl The results will be aggregated to arrive at one reported value (e.g., Number of Participants with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment)

IPD SHARING:
Plan to Share IPD: Undecided